CLINICAL TRIAL: NCT02298491
Title: Clinical Biomarkers of Disease Activity and Treatment Responses in Patients With CNS Sarcoidosis Treated With H.P. Acthar Gel
Brief Title: CNS Sarcoidosis and Acthar Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Horea Rus, Professor of Neurology, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00062490
Record Dates: First submitted 2014-11-14; First posted 2014-11-24 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: CNS Sarcoidosis
MeSH Terms: interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- H.P. Acthar Gel (Experimental)
  Interventions: Drug: H.P. Acthar Gel

INTERVENTIONS:
Drug: H.P. Acthar Gel — 80 IU subcutaneously daily for 10 days then followed by 80 IU subcutaneously three times per week through Month 12
  Other Names: ACTH

SUMMARY:
The purpose of this study is to see if treatment with H.P. Acthar® Gel will result in the improvement and long-term stabilization of clinical and radiographic abnormalities that occur in patients with CNS sarcoidosis. In addition, it will also look at whether treatment will be also associated with improvement in measures of quality of life. The treatment of CNS sarcoidosis involves the use of either corticosteroids such as prednisone or potent immunosuppressive agents such as methotrexate, both which can induce severe long term side effects. The adverse effects of steroids may be avoided by treatment with adrenocorticotropic hormone (ACTH), which is available for patient use as H.P. Acthar® Gel. The efficacies of H.P. Acthar® Gel in the treatment of CNS sarcoidosis and the impact on quality of life have not been previously studied. In addition, little is known regarding the expression of immune markers in CNS sarcoidosis and the association of such markers with disease activity and response to treatment.

DETAILED DESCRIPTION:
Sarcoidosis is a chronic and frequently progressive systemic disease that affects the central nervous system (CNS) in approximately 5% of patients. The hallmark of the disease is the development of chronic inflammation with formation of non-caseating granulomas that can involve the brain parenchyma and meninges and appear as contrast-enhancing mass lesions on magnetic resonance imaging. The granulomas are primarily comprised of proinflammatory T cells (Th1 cells and Th17 cells) and macrophages which accumulate during the early stages of granuloma formation. The inflammation that is generated by these cells is modulated by anti-inflammatory responses mediated by Th2 cells and regulatory T (Treg) cells that later appear and populate the outer regions of the granuloma. The presence of Treg cells are of particular interest since these cell are also detected in high numbers in peripheral blood and the immune suppression that results may underlie the occurrence of anergy in patients with the disease. The treatment of CNS sarcoidosis involves the use of either corticosteroids or potent immunosuppressive agents, both which can induce severe long-term side effects. The adverse effects of steroids may be avoided by treatment with adrenocorticotropic hormone (ACTH), which is available for patient use as H.P. Acthar® Gel. The efficacy of H.P. Acthar® Gel in the treatment of CNS sarcoidosis and the impact on quality of life have not been previously examined. In addition, little is known regarding the expression of immune markers in CNS sarcoidosis and the association of such markers with disease activity and response to treatment. These issues, therefore, will be explored in the context of this proposal.

ELIGIBILITY:
Inclusion Criteria:

* A highly probable diagnosis of sarcoidosis, as determined using the World Association for Sarcoidosis and Other Granulomatous Disorders (WASOG) Sarcoidosis Organ Assessment Instrument (Judson et al., 2014), with involvement not limited to the central nervous system.
* At the time of enrollment, a history of clinical deterioration based on the development of new symptoms or worsening previously present symptoms with confirmation by clinical examination and objective clinical testing.
* If on steroids, on a stable dose of the medication for at least 3 months.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-05; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horea Rus, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Background] Agostini C, Meneghin A, Semenzato G. T-lymphocytes and cytokines in sarcoidosis. Curr Opin Pulm Med. 2002 Sep;8(5):435-40. doi: 10.1097/00063198-200209000-00016. PMID 12172449
- [Background] Arnason BG, Berkovich R, Catania A, Lisak RP, Zaidi M. Mechanisms of action of adrenocorticotropic hormone and other melanocortins relevant to the clinical management of patients with multiple sclerosis. Mult Scler. 2013 Feb;19(2):130-6. doi: 10.1177/1352458512458844. Epub 2012 Oct 3. PMID 23034287
- [Background] Co DO, Hogan LH, Il-Kim S, Sandor M. T cell contributions to the different phases of granuloma formation. Immunol Lett. 2004 Mar 29;92(1-2):135-42. doi: 10.1016/j.imlet.2003.11.023. PMID 15081537
- [Background] Judson MA, Costabel U, Drent M, Wells A, Maier L, Koth L, Shigemitsu H, Culver DA, Gelfand J, Valeyre D, Sweiss N, Crouser E, Morgenthau AS, Lower EE, Azuma A, Ishihara M, Morimoto S, Tetsuo Yamaguchi T, Shijubo N, Grutters JC, Rosenbach M, Li HP, Rottoli P, Inoue Y, Prasse A, Baughman RP, Organ Assessment Instrument Investigators TW. The WASOG Sarcoidosis Organ Assessment Instrument: An update of a previous clinical tool. Sarcoidosis Vasc Diffuse Lung Dis. 2014 Apr 18;31(1):19-27. PMID 24751450
- [Background] Miller DH, Kendall BE, Barter S, Johnson G, MacManus DG, Logsdail SJ, Ormerod IE, McDonald WI. Magnetic resonance imaging in central nervous system sarcoidosis. Neurology. 1988 Mar;38(3):378-83. doi: 10.1212/wnl.38.3.378. PMID 3347340
- [Background] Miyara M, Amoura Z, Parizot C, Badoual C, Dorgham K, Trad S, Kambouchner M, Valeyre D, Chapelon-Abric C, Debre P, Piette JC, Gorochov G. The immune paradox of sarcoidosis and regulatory T cells. J Exp Med. 2006 Feb 20;203(2):359-70. doi: 10.1084/jem.20050648. Epub 2006 Jan 23. PMID 16432251
- [Background] Moller DR. Treatment of sarcoidosis -- from a basic science point of view. J Intern Med. 2003 Jan;253(1):31-40. doi: 10.1046/j.1365-2796.2003.01075.x. PMID 12588536
- [Background] Royal W 3rd, Mia Y, Li H, Naunton K. Peripheral blood regulatory T cell measurements correlate with serum vitamin D levels in patients with multiple sclerosis. J Neuroimmunol. 2009 Aug 18;213(1-2):135-41. doi: 10.1016/j.jneuroim.2009.05.012. Epub 2009 Jun 17. PMID 19539379
- [Background] Shi C, Pamer EG. Monocyte recruitment during infection and inflammation. Nat Rev Immunol. 2011 Oct 10;11(11):762-74. doi: 10.1038/nri3070. PMID 21984070
- [Background] Stern BJ, Aksamit A, Clifford D, Scott TF; Neurosarcoidosis Study Group. Neurologic presentations of sarcoidosis. Neurol Clin. 2010 Feb;28(1):185-98. doi: 10.1016/j.ncl.2009.09.012. PMID 19932381
- [Background] Stern BJ, Krumholz A, Johns C, Scott P, Nissim J. Sarcoidosis and its neurological manifestations. Arch Neurol. 1985 Sep;42(9):909-17. doi: 10.1001/archneur.1985.04060080095022. PMID 3896208

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | H.P. Acthar Gel
Started | 4
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 46.3 [40 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Lesions
Description: Total number of lesions assessed at 1 year
Time Frame: 1 year
Measure: Number; unit: lesions
Arm/Group | H.P. Acthar Gel
Number analyzed (Participants) | 3
lesions | 5

2. Secondary Outcome: Quality of Life Measures
Description: Change in Patient Determined Disease Steps (PDDS), Montreal Cognitive Assessment (MoCA), Symbol-Digit Modalities Test (SDMT), Short Form -36 Health Survey (SF-36), Work Productivity and Activities Impairment -General Health (WPAI-GH) and Beck Depression Inventory-II (BDI-II) at 4 weeks, 6 months and 12 months relative to baseline
Time Frame: 4 weeks, 6 months and 12 months
Reporting Status: Not Posted, anticipated posting 2021-11

3. Secondary Outcome: Quality of Life Measure
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) scores at 4 weeks and change in TSQM scores at 6 months and 12 months versus baseline
Time Frame: 6 months and 12 months
Reporting Status: Not Posted, anticipated posting 2021-11

4. Other Pre Specified Outcome: Serum and Cerebrospinal Fluid Immune Markers
Description: Change in levels of serum and cerebrospinal fluid immune markers at 4 weeks, 6 months and 12 months versus baseline
Time Frame: 4 weeks, 6 months and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | H.P. Acthar Gel
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2014-07-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT02298491/Prot_000.pdf